CLINICAL TRIAL: NCT04194554
Title: A Multi-Center Trial of Androgen Suppression With Abiraterone aCetate, LEuprolide, PARP Inhibition and Stereotactic Body Radiotherapy (ASCLEPIuS): A Phase I/2 Trial in High Risk and Node Positive Prostate Cancer
Brief Title: A Multi-Center Trial of Androgen Suppression With Abiraterone Acetate, Leuprolide, PARP Inhibition and Stereotactic Body Radiotherapy in Prostate Cancer
Acronym: ASCLEPIuS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2019.117; HUM00167325 (Other: University of Michigan)
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — niraparib; Leuprolide; Abiraterone Acetate; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Time to Event Continual Reassessment Method (TITE-CRM) dose-finding clinical trial design.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Niraparid Dose Escalation (Experimental): Dose Level 1: 100 mg PO daily of Niraparib but held for 5 days (+/- 2 days) prior to RT, during SBRT, and 5 days (+/- 2 days) after last fraction of SBRT
  Dose Level 2: 200 mg PO daily of Niraparib but held for 5 days (+/- 2 days) prior to RT, during SBRT, and 5 days (+/- 2 days) after last fraction of SBRT
  Dose Level 3: 200 mg PO daily of Niraparib without breaks during SBRT until completion of 6 cycles.
  Interventions: Drug: Niraparib; Drug: Leuprolide; Drug: Abiraterone Acetate; Radiation: Stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Drug: Niraparib — given PO per dose escalation schedule
Drug: Leuprolide — 22.5 mg q3 month
Drug: Abiraterone Acetate — 1000 mg daily
Radiation: Stereotactic body radiotherapy (SBRT) — 5-6 fraction SBRT (total dose: 37.5-40 Gy)
  Other Names: Ultra-hypofractionated radiotherapy

SUMMARY:
The purpose of this study is to establish the maximum tolerable dose of niraparib when combined with prostate stereotactic body radiotherapy (SBRT), abiraterone, leuprolide, and prednisone (the phase 1 portion of the study) and determine 3-year biochemical PSA recurrence free-survival with this treatment approach (the phase 2 portion of the study).

ELIGIBILITY:
Inclusion Criteria

1. Pathologic biopsy proven adenocarcinoma of the prostate
2. At least one of the following criteria:

   * cN1 on conventional or PET imaging
   * Grade group 5
   * Grade group 4
   * Grade group 3 and PSA ≥20 ng/mL
   * High probability of Radiographic T3 on MRI AND Grade group ≥2
   * Grade Group 3 AND PSA ≥10 ng/mL AND ≥50% positive biopsy cores
3. Age ≥ 18
4. ECOG < 1
5. Adequate organ and marrow function as defined per protocol.
6. Use of highly effective contraception (e.g. condoms) for the duration of treatment and a minimum of 120 days thereafter. Men must also agree not to donate sperm for the duration of the study participation, and for at least 120 days thereafter.
7. International Prostate Symptoms Score (IPSS) ≤ 20
8. Medically fit for treatment and agreeable to follow-up
9. Ability to understand and the willingness to sign a written informed consent
10. Tissue available for MiOncoSeq testing to assign DNA repair deficiency status

Exclusion Criteria

1. Clinical or radiographic evidence of distant metastatic disease by CT/bone scan
2. Clinical or radiographic evidence of high probability of clinical T4 disease
3. Prostate gland size >80 cc measured by ultrasound or MRI
4. Prominent median lobe assessed by treating physician
5. Lack of tissue from biopsy to be sent for correlative studies
6. Any prior treatment for prostate cancer (incudes history of TURP within 5 years of enrollment, chemotherapy, radiation therapy, or anti-androgen therapy)
7. Prohibited within 30 days prior to administration to study treatment: spironolactone and other investigational drug therapies.
8. Prohibited 3 months before participant registration and during administration of study treatment: non-steroidal anti-androgens (e.g., bicalutamide, flutamide, nilutamide), steroidal antiandrogens (megestrol acetate, cyproterone acetate), oral ketoconazole, chemotherapy, immunotherapy, estrogens, radiopharmaceuticals.
9. History of prior pelvic radiation therapy
10. Concurrent treatment with strong CYP3A4 inducers such as phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital
11. Enrollment concurrently in another investigational drug study within 1 month of registration
12. History of another active malignancy within the previous 3 years except for adequately treated skin cancer or superficial bladder cancer
13. History of or active Crohn's disease or ulcerative colitis
14. Contraindication to or inability to tolerate MRIs
15. Patients with severe depression
16. Uncontrolled diabetes or known HbA1c>10
17. Any gastrointestinal disorder affecting absorption
18. Active pituitary or adrenal dysfunction
19. Patients with significant cardiovascular disease potentially including severe / unstable angina, recent history of myocardial infarction, clinically significant heart failure, cerebrovascular disease, venous thromboembolic events, clinically significant arrhythmias)
20. Uncontrolled hypertension with persistently elevated systolic blood pressure >160 mmgHg or diastolic blood pressure >100 mmHg despite anti-hypertensive agents.
21. Prolonged QTc >450 ms or any ECG changes that interfere with QT interval interpretation
22. Major surgery within 1 month of registration
23. History of myelodysplastic syndrome or leukemia
24. A known hypersensitivity to niraparib, abiraterone acetate, leuprolide, and/or prednisone
25. Active infection or other medical condition that would be a contraindication to prednisone use
26. Patients with known active hepatitis or chronic liver disease including cirrhosis
27. Any condition that in the opinion of the investigator would preclude participation in this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (Phase 1) | Up to 112 days after initial dose of niraparib
  The proportion of patients at each dose level with dose-limiting toxicity (DLT), defined as any treatment related grade 3-5 adverse event experienced within the first 4 treatment cycles (112 days), assessed per NCI's CTCAE version 5.0.
Proportion of patients experiencing biochemical failure | Up to 3 years after first dose of niraparib
  Change in PSA level from the beginning of study treatment for up to 3 years later will determine the biochemical failure rate. Biochemical failure will be defined using the Phoenix definition of the PSA nadir + 2 ng/mL.

SECONDARY OUTCOMES:
Change in health related quality of life | From baseline up to 3 years after last dose of niraparib
  Assessed via EPIC-26 questionnaire
Proportion of patients with undetectable post-treatment PSA | Measured during the end of the 6th cycle of therapy (during week 24 +/- 7 days)
  Undetectable PSA will be defined as a PSA ≤0.1 ng/mL.
Proportion of patients with distant metastases | Up to 5 years after first dose of niraparib
  Distant metastases will be defined as any clinical or radiographic evidence of lymph node, bone, or visceral involvement of prostate cancer.
Prostate cancer specific survival | Up to 5 years after first dose of niraparib
  Prostate cancer specific survival will be defined as the duration of time from the start of treatment to death attributable to prostate cancer. Patients who have not died or die of non-prostate cancer related causes will be censored at the last known follow-up or date of death, respectively. Summarized using cumulative incidence or Kaplan-Meier curves as appropriate.
Overall survival | Up to 5 years after first dose of niraparib
  Overall survival (OS) will be defined as the duration of time from the start of treatment to death from any cause. Patients who have not died will be censored at the last known follow-up.Summarized using cumulative incidence or Kaplan-Meier curves as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Spratt, M.D., Study Chair — Case Western Reserve University - Seidman Comprehensive Cancer Center; William Jackson, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (6):
- United States (6):
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cornell University, New York, New York
  - Weill Cornell Medicine, New York, New York
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data that may be shared will only include individual participant data that underlie the results reported publicly in ClinicalTrials.gov or published articles, after deidentification (text, tables, figures, appendices).
Supporting Information: Study Protocol
Time Frame: The time frame for data sharing will begin 12 months after the initial publication and continue until 36 months after publication in ClinicalTrials.gov.
Access Criteria: Once the final results of the trial have been reported parties interested in accessing the data should contact the trial PI (Dr. Daniel Spratt) to discuss any potential data sharing requests. An analysis plan is required and intended use of the data must be disclosed. Only de-identified data may be shared and all agreements must comply with current policies of both parties to share data.